CLINICAL TRIAL: NCT03639805
Title: Effect of a Music Therapy Program on Vaso-occlusive Crisis Pain in Sickle Cell Disease Patients: A Pilot Study
Brief Title: Music Therapy in Sickle Cell Disease Vaso-occlusive Crisis
Acronym: MUSICODREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K171205J
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Vaso-occlusive Crisis
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non interventional arm (Active Comparator): Standard Of Care
  Interventions: Other: standard care of vaso-occlusive crises
- interventional arm (Experimental): Standard of Care + music therapy program MUSIC CARE®
  Interventions: Other: Music therapy program MUSIC CARE® + standard care

INTERVENTIONS:
Other: Music therapy program MUSIC CARE® + standard care — Administration of a specific music therapy program (U method) delivered through headphones from an iPad, under the direction of trained nurses. The program will be proposed 3 times a day and will last 20 minutes at each session.
  Arms: interventional arm
Other: standard care of vaso-occlusive crises — administration of standard care only
  Arms: non interventional arm

SUMMARY:
Treatment of painful vaso-occlusive crises, the most common manifestation of sickle cell disease, is notoriously limited. vaso-occlusive crises pain is multifactorial with a psychological component. The hypothesis is that the music therapy program MUSIC CARE® can help alleviate severe vaso-occlusive crises pain in synergy with traditional treatment in sickle cell disease patients. The main objective of this prospective, randomized, open label study is to test the effect of the music therapy program MUSIC CARE® on daily mean morphine consumption during the 3 first days of hospitalisation for severe vaso-occlusive crises.

DETAILED DESCRIPTION:
Sickle cell disease, the most frequent monogenic disease in France and in the world, is induced by a mutation in the β-globin chain of hemoglobin with production of hemoglobin S. The course of the disease is characterized by very painful, for which treatment is notoriously limited. vaso-occlusive crises pain is multifactorial with biological and psychological components. A few studies suggest a beneficial effect of relaxation techniques in the management of Sickle cell disease pain. MUSIC CARE® is a novative music therapy program which proved efficient in different models of acute or chronic pain. the hypothesis is that this program can help alleviate severe pain in synergy with traditional treatment in SS Sickle cell disease patients, via a dual biological and psychological effect. The main objective of this prospective, randomized, open label study is to test the effect of the music therapy program MUSIC CARE® on daily mean morphine consumption during the 3 first days of hospitalisation for severe vaso-occlusive crises in adult SS Sickle cell disease patients. Secondary outcomes will include mean daily Visual Analogic Scale during the first 3 days of hospitalization for severe vaso-occlusive crises, acute complications of vaso-occlusive crises, duration of severe vaso-occlusive crises and of hospitalization, Hospital Anxiety and Depression Scale.

20 patients will be included in each group for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* patients with homozygous Sickle Cell Disease (HbSS,or HbSß0) confirmed by laboratory center
* hospitalized for severe vaso-occlusive crisis
* Visual Analogic Scale≥6 at entry
* able to speak and write French
* Patient in physical and clinical capacity of consent (signature of the informed consent of the patient or in the presence of a third party)
* affiliated to a social insurance; not subject to a legal protection

Exclusion Criteria:

* other hemoglobinopathy
* pregnancy or post-scriptum (40 days after labor)
* antecedent of Reflex Epilepsies
* major hypoacusia
* Patients already engaged in a therapeutic protocol or in the period of exclusion after a previous interventional research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-04-28 (Estimated); Study Completion 2020-04-28 (Estimated)

PRIMARY OUTCOMES:
Daily mean morphine consumption during the first 3 days of hospitalization for severe vaso-occlusive crises | End of the third day of hospitalization for severe vaso-occlusive crises
  The total morphine consumption will be calculated for the first 3 days of hospitalization by a doctor, and a mean daily consumption will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain LE JEUNE, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Avicenne University Hospital, Bobigny, France